CLINICAL TRIAL: NCT01785862
Title: Study of Efficacy and Safety of V0498 Versus Placebo in Acute Sore Throat Pain.
Brief Title: Ibuprofen Lozenge in Acute Sore Throat Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V00498 TA 3 01; 2012-004423-20 (EudraCT Number)
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Acute Sore Throat Pain
Keywords: sore throat pain; tonsillopharyngitis; upper respiratory tract infection
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Drug (Experimental): V0498, Ibuprofen 25 mg
  Interventions: Drug: Ibuprofen 25 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen 25 mg — Lozenge, Oromucosal administration
  Arms: Drug
Drug: Placebo — Lozenge matching V0498 lozenge, Oromucosal administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of repeated doses of a low dosage of oromucosal Ibuprofen form (lozenge) versus placebo in patients suffering from acute sore throat pain.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged at least 18 years old
* patient with an acute sore throat

Exclusion Criteria:

* Severe respiratory tract infection (pneumonia, bronchitis or laryngitis)
* Oro-pharyngeal paresthesia or mycosis
* Severely traumatised and/or very severe oromucosal inflammation
* Tonsillopharyngectomy
* Peritonsillar abscess
* Hypersensitivity to ibuprofen or other NonSteroidal Anti-Inflammatory Drugs (NSAIDs) (including bronchospasm) or to excipients
* Long term use (≥ 3 times per week within the last month or regular intake within the last 3 months before randomisation) of antiinflammatory drugs- Any long-acting or slow release analgesic intake including NonSteroidal Anti-Inflammatory Drugs (NSAIDs)within 24 hours before randomisation (e.g. piroxicam or naproxen)
* Any anti-inflammatory drugs intake by systemic route within 12 hours before randomisation
* Any paracetamol intake within 6 hours before randomisation
* Any cold medication (decongestant, antihistamine, expectorant, antitussive) within 6 hours before randomisation
* Any topical throat medication intake containing or not a local oral anaesthetic such as lozenge, spray, mouth rinse within 4 hours before randomisation
* Heavy smokers (>20 cigarettes/day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Total Pain relief over 2 hours | 0-2 hours post-dose
  Total Pain Relief (TOTPAR) assessed on a 7-point rating scale called the Sore Throat Relief Scale (STRS) over 120min after the start of sucking of 1st study drug administered

CONTACTS AND LOCATIONS:
Locations (14):
- Gières, France
- Erfurt, Germany
- Latvia (10):
  - Balvi
  - Daugavpils
  - Jelgava
  - Jēkabpils
  - Kuldīga
  - Liepāja
  - Ogre
  - Ogres Municipality
  - Riga
  - Saldus
- United Kingdom (2):
  - Cardiff
  - Glasgow

REFERENCES:
- [Derived] Bouroubi A, Donazzolo Y, Donath F, Eccles R, Russo M, Harambillet N, Gautier S, Montagne A. Pain relief of sore throat with a new anti-inflammatory throat lozenge, ibuprofen 25 mg: A randomised, double-blind, placebo-controlled, international phase III study. Int J Clin Pract. 2017 Sep;71(9). doi: 10.1111/ijcp.12961. Epub 2017 Sep 4. PMID 28869722